CLINICAL TRIAL: NCT00167245
Title: A Phase II, Randomized, Double-blind, Placebo-Controlled, Pilot Trial of Topiramate for Alcohol and Comorbid Cocaine Dependence
Brief Title: Topiramate for Alcohol and Cocaine Dependence
Acronym: TOP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyle Kampman (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Kyle Kampman, Sponsor-Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 801385; R01AA014657 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2019-07

CONDITIONS: Alcoholism; Cocaine Dependence
Keywords: Topiramate; alcoholism; cocaine dependence
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): topiramate capsules dose titrated up to 300 mg daily
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): placebo capsules identical in appearance to the topiramate capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Topiramate — 300mg/day for 13 weeks
  Other Names: topamax
  Arms: Topiramate
Drug: placebo — placebo pills
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to test the effectiveness of topiramate for the treatment of combined alcohol and cocaine dependence. Topiramate is approved for the treatment of seizures. It has not been proven to be effective for the treatment of alcohol or cocaine dependence.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of 300 mg/day of topiramate for the treatment of 200 treatment-seeking alcohol dependent outpatients with comorbid cocaine dependence in a double-blind, placebo-controlled 14-week trial, with a 6-month follow-up (3 months after completing medications).

ELIGIBILITY:
Inclusion Criteria:

* Male and females, 18 years or older.
* Meets DSM(Diagnostic and Statistical Manual)-IV criteria for current diagnoses of cocaine and alcohol dependence, determined by the SCID (Structured Clinical Interview for the DSM)-IV.
* In the past 30 days, used no less than $200-worth of cocaine and meets the following drinking criteria as measured by the Timeline Followback (TLFB) (Sobell and Sobell, 1995) a. drank within 30 days of intake day, b. reports a minimum of 48 standard alcoholic drinks (avg. 12 drinks/wk) in a consecutive 30-day period over the 90-day period prior to starting intake (i.e., a minimum of 40% days drinking), and c. has 2 or more days of heavy drinking (defined as 5 or more drinks per day in males and 4 or more drinks per day in females) in this same pre-treatment period.
* Two consecutive days of abstinence from cocaine and alcohol, determined by self-reports and confirmed by negative urine toxicology screens, a negative breathalyzer tests, and collateral report, a Clinical Institute Withdrawal Scale for Alcohol (CIWA-AR) (Sullivan et al., 1989) score below eight,. Subjects will be encouraged to achieve 3 consecutive days of abstinence, however, subjects who have achieved 2 consecutive days of abstinence will be included with the approval of the principal investigator. We anticipate that these subjects will comprise less than 5% of total enrolled subjects. Subjects will be given 2 additional weeks beyond the screening week to attain the appropriate period of cocaine and alcohol abstinence prior to randomization.
* Lives a commutable distance from the Treatment Research Center (TRC) and agrees to attend all research visits including follow-up visits.
* Speaks, understands, and prints in English.

Exclusion Criteria:

* Abstinent from cocaine or alcohol for 30 consecutive days prior to signing consent form.
* Meets DSM-IV criteria for dependence on any substance other than cocaine and alcohol (except nicotine and cannabis), determined by the SCID.
* Needs treatment with any psychoactive medications including any anti-seizure medications (with the exception of Benadryl used sparingly, if necessary, for sleep).
* Current use of phenytoin or any drug of similar class.
* Meets DSM-IV criteria for schizophrenia or any psychotic disorder, or organic mental disorder. Subject meets current DSM-IV diagnosis of any other clinically significant psychiatric disorder that will interfere with study participation.
* Has evidence of a history of significant hematological, pulmonary, endocrine, cardiovascular, renal or gastrointestinal disease.
* Severe physical or medical illnesses such as AIDS, active hepatitis, significant hepatocellular injury as evidenced by elevated bilirubin levels (>1.3), or elevated levels (over 3.5x normal) of aspartate aminotransferase (AST), and serum glutamic-pyruvic transaminase (SGPT) after the required 3 days of abstinence, or severe renal disease, severe respiratory diseases or severe diarrhea with resulting metabolic acidosis, serum bicarbonate (< 20 milliequivalent (mEq)/L)
* History of epilepsy or seizure disorder.
* Use of an investigational medication in the 30 days prior to randomization.
* History of nephrolithiasis (kidney stones).
* History of hypersensitivity to topiramate.
* Is female and tests positive on a pregnancy test, is contemplating pregnancy in the next 6 months, is nursing, or is not using an effective contraceptive method (if relevant). Acceptable methods of contraception include barrier methods (diaphragm or condom with spermicide, intrauterine progesterone contraceptive system, levonorgestrel implant, and medroxyprogesterone acetate contraceptive injection).
* Current use of a carbonic anhydrase inhibitor.
* A history of glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2004-09; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Kampman, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study began on 11/1/2004 and ended five years later in November 2009. Participants were treatment-seeking cocaine and alcohol users recruited at the UPenn Treatment Research Center.
Groups:
- Topiramate: topiramate
  Topiramate : 300mg/day for 13 weeks
- Placebo: placebo : placebo pills
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 83 | 87
Completed | 54 | 46
Not Completed | 29 | 41
Not completed — Lost to Follow-up | 20 | 31
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Incarcerated | 3 | 2
Not completed — Drowsy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: topiramate
  Topiramate : 300mg/day for 13 weeks
- Group 2: placebo : placebo pills
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 83 | 87 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 87 | 170
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (7.0) | 43 (8.0) | 44 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 65 | 69 | 134
Region of Enrollment [Number; unit: participants]
  United States | 83 | 87 | 170

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Abstinent From Cocaine During Last 3 Weeks of 13 Week Trial
Description: Samples were analyzed for benzoylecgonine by fluorescent polarization assay. Samples containing equal to or greater than 300 ng/ml of benzoylecgonine were considered to be positive for cocaine.
Time Frame: Last 3 weeks of 13 week trial
Measure: Number; unit: Percent of participants
Groups:
- Topirmate: topiramate
  Topiramate : 300mg/day for 13 weeks
Arm/Group | Topirmate | Placebo
Number analyzed (Participants) | 83 | 87
Percent of participants | 17 | 6
Statistical Analysis 1: Comparison: Topirmate vs Placebo; Test type: Superiority; p = 0.01, Chi-squared

2. Primary Outcome: Number of Heavy Drinking Days
Description: Heavy drinking days, defined as more than 4 standard drinks for men and 3 standard drinks for women
Time Frame: 13 weeks
Measure: Mean (Standard Error); unit: number of heavy drinking days
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 54 | 46
number of heavy drinking days | 5.21 (.58) | 6.10 (.61)
Statistical Analysis 1: Comparison: Topiramate vs Placebo; Test type: Superiority or Other; p = 0.45, Generalized Estimating Equations

3. Secondary Outcome: Cocaine Withdrawal Symptoms Measured by Cocaine Selective Severity Assessment.
Description: Total cssa score at the end of the medication phase of the trial. The CSSA is a measure of cocaine withdrawal severity. The minimum score is 0 the maximum score is 119. Higher score means more severe cocaine withdrawal symptoms
Time Frame: 13 weeks
Population: Subjects present during the last week of the trial
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group 1: topiramate
  Topiramate: 300mg/day for 13 weeks
- Group 2: placebo: placebo pills
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 52 | 47
score on a scale | 9.9 (9.5) | 8.4 (8.8)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = 0.4, t-test, 2 sided; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-2.1 to 5.2]

4. Secondary Outcome: The Penn Alcohol Craving Scale
Description: This Scale measures alcohol craving. The maximum score is 30, the minimum score is 0. Higher scores are indicative of more severe alcohol craving.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 83 | 87
score on a scale | 7.90 (6.86) | 9.29 (6.48)

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: adverse events queried at each visit
Arm/Group | Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/87
Other Adverse Events (participants affected / at risk) | 46/83 | 24/87
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=83) | Placebo (N=87)
Sedation (General disorders) | 17 | 15
Paresthesias (Skin and subcutaneous tissue disorders) | 17 | 3
Headache (General disorders) | 6 | 3
Dry Mouth (General disorders) | 6 | 3

LIMITATIONS AND CAVEATS:
The total number of subjects was relatively small and thus the results should be considered preliminary. The study drop-out rate was formidable, though it was comparable with most trials involving cocaine-dependent patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes